CLINICAL TRIAL: NCT06776835
Title: Screening of Small Non-coding RNAs as an Auxiliary Diagnostic Biomarker for Gastric Cancer and Exploring Its Correlation With Prognostic Diagnosis
Brief Title: Screening of Small Non-coding RNAs as an Auxiliary Diagnostic Biomarker for Gastric Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-L166
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gastric cancer cases from medical centers in China: Measurement of levels of circulating small non-coding RNAs
  Interventions: Diagnostic Test: Analysis of relative quantitative of small non-coding RNAs
- Controls from medical centers in China: Measurement of levels of circulating small non-coding RNAs
  Interventions: Diagnostic Test: Analysis of relative quantitative of small non-coding RNAs

INTERVENTIONS:
Diagnostic Test: Analysis of relative quantitative of small non-coding RNAs — Each participant was enrolled to assess the of relative quantitative of small non-coding RNAs

SUMMARY:
Gastric cancer is one of the most common malignancies of the gastrointestinal system, especially in East Asia. A host of patients are diagnosed with GC at the late stage, leading to poor patient prognosis. Therefore, there is a strong demand to develop new biomarkers to detect this tumor early. Small non-coding RNA species include microRNA (miRNA), PIWI-interacting RNA (piRNA), small interfering RNA (siRNA), tRNA-derived small RNA (tsRNA), etc. It has been demonstrated that small non-coding RNAs are involved in gastric cancer cell proliferation, metastasis, progression and survival. Hence, it is considered as an auxiliary diagnostic biomarker for gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignancies of the gastrointestinal system, especially in East Asia. A host of patients are diagnosed with GC at the late stage, leading to poor patient prognosis. Therefore, there is a strong demand to develop new biomarkers to detect this tumor early.

Small non-coding RNA species include microRNA (miRNA), PIWI-interacting RNA (piRNA), small interfering RNA (siRNA), tRNA-derived small RNA (tsRNA), etc. It has been demonstrated by previous scientific researches that small non-coding RNAs are involved in gastric cancer cell proliferation, metastasis, progression and survival. Hence, it is considered as a new biomarker panel for gastric cancer.

The purpose of the present clinical trail is to explore the correlation between small non-coding RNAs panel and early gastric cancer, and to elucidate the possibility of small non-coding RNAs panel as a biomarker for gastric cancer. Verify the experimental purpose by monitoring the relative quantification of small non-coding RNAs panel through high-throughput sequencing and qRT PCR technology.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old and ≤ 85 years old
* Histologically confirmed gastric cancer

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AFFILIATED HOSPITAL OF NANTONG UNIVERSITY
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Analysis of relative quantitative of small non-coding RNAs | an average of 2 years
  Relative quantitative of small non-coding RNAs are detected by quantitative RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided